CLINICAL TRIAL: NCT01899807
Title: Cranial Reconstruction With Patient-specific Titanium Mesh/Mosaic-designed Calcium Phosphate-implant - A Multi Center Center, Single Arm, Non-comparative Prospective Case Series
Brief Title: Bone Reconstruction of the Skull Using a Metal Ceramic Implant After Previously Failed Reconstruction
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Karolinska University Hospital (Other)
Responsible Party: Principal Investigator, Dr. Kalle Lundgren, MD, PhD, Karolinska University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OQ-CR-001
Record Dates: First submitted 2013-07-02; First posted 2013-07-15 (Estimated); Last update posted 2015-03-31 (Estimated); Status verified 2015-03

CONDITIONS: Defect of Skull Ossification; Other Specified Skull or Face Bone Anomaly; Cranial Dysostosis Nec; Hemicraniectomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Single Arm (Other)
  Interventions: Device: OssDsign AB

INTERVENTIONS:
Device: OssDsign AB

SUMMARY:
The purpose of this study is to evaluate a new ceramic metal bone graft substitute for hemi craniectomies. The frequency of infections and rupture of skin will be studied, which is a reoccurring problem with currently used bone graft substitutes in this subject population. In addition, the quality of life before and after implantation will be evaluated as well as the bone regeneration around implant.

ELIGIBILITY:
Inclusion Criteria:

* Obtained informed consent.
* Males or females, ≥18 years of age
* Subject with cranial defect size > 25 cm2.
* History of previous cranial implant failure and where the latest cranial reconstruction failed within 12 months. (This means that the patient demonstrates a non-reconstructed cranial defect after removal of implant or exhibit an implant failure, e.g. local infection and/or protrusion through the skin.)
* Willing and able to comply with all study procedures and restrictions.
* The 5 subjects participating in bone regeneration analysis (PET/CT scans) has to be 50 years or older

Exclusion Criteria:

* Malignancy adjacent to the reconstruction area, including brain and calvaria, with on-going or planned surgical intervention.
* Pregnant or nursing women.

Exclusion criteria during surgery, if applicable:

Perioperative appearance of previously not identified tumor or infection in the reconstruction area.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2013-06; Primary Completion 2016-03 (Estimated); Study Completion 2016-03 (Estimated)

PRIMARY OUTCOMES:
Rate of adverse events | From the date of intervention up to 12 months post intervention
  The primary endpoint, rate of adverse events, will be measured by clinical evidence of infection and/or manifested rupture of skin around the implant, within 12 months, that necessitates explantation.

SECONDARY OUTCOMES:
Percentage subjects with an adverse event | From the date of intervention up to 14 days, 3 months, 6 months follow-up
Quality of life scores | Assessed during the 3 month- and 12 month follow-up visit post intervention, compared to the screening visit: 3-0 weeks prior to intervention
  SF-12 and EQ5D 3L will be used
PET/CT analysis with bone tracer, confirms bone regeneration activity within the reconstruction area | The PET/CT scan will be taken at 12 months post intervention and it will be compared with 2 weeks post intervention
  The bone tracer (18 F fluoride) will be used to measure bone regeneration.
Subject mean MOCA | 3 months and 12 months follow-up compared to baseline
  Subject cognitive impairment is measured by Montreal Cognitive Assessment (MOCA) (the subject will be given a score after completing the assessment)

OTHER OUTCOMES:
Health economy variables | 3 months and 12 months post intervention compared to baseline visit: 3-0 weeks pre intervention
  Mean number of hospital days, hospital visits, mean time to adverse event and lost work days related to the study treatment will be counted.

CONTACTS AND LOCATIONS:
Overall Officials: Lars Kihlström, MD, MBA, Principal Investigator — Department of Neurosurgery, Karolinska University Hospital; Kalle Lundgren, MD, PhD, Principal Investigator — Karolinska University Hospital
Locations (2):
- Sweden (2):
  - Dept. of Neurosurgery, Sahlgrenska University Hospital, Gothenburg
  - Dept. of Neurosurgery, Karolinska Universitetssjukhuset, Stockholm